CLINICAL TRIAL: NCT02232217
Title: Cognitive Behavioral Treatment for Improving Sleep in Overweight and Obese Youth
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Florida (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: IRB201400307-N; R21HL121432 (NIH); NIH NHLBI [pending] (Other: R21HD11680545)
Record Dates: First submitted 2014-09-02; First posted 2014-09-05 (Estimated); Last update posted 2018-05-11 (Actual); Status verified 2018-05

CONDITIONS: Sleep
Keywords: Children; Sleep; Obesity
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Cognitive Behavior Therapy Sleep (Experimental): Children in this arm will receive instructions on the use of 'coping thoughts.' Common elements across the CBTcs sessions include reviewing progress, setting goals for change, problem solving to address challenges/barriers, and reinforcing progress
  Interventions: Behavioral: Cognitive Behavior Therapy Sleep
- Education Control (Active Comparator): Children in this arm will receive sleep and dietary education, as well as general coping strategies and controls for staff attention and seasonal effects that could influence changes in sleep and health outcomes.
  Interventions: Other: Education Control

INTERVENTIONS:
Behavioral: Cognitive Behavior Therapy Sleep — Children in this arm will receive instructions on the use of 'coping thoughts.' Common elements across the CBTcs sessions include reviewing progress, setting goals for change, problem solving to address challenges/barriers, and reinforcing progress
  Other Names: CBTcs
  Arms: Cognitive Behavior Therapy Sleep
Other: Education Control — Children in this arm will receive sleep and dietary education, as well as general coping strategies and controls for staff attention and seasonal effects that could influence changes in sleep and health outcomes.
  Other Names: EC
  Arms: Education Control

SUMMARY:
The purpose of this study is to conduct a randomized controlled trial (RCT) to evaluate the efficacy of brief cognitive behavioral treatment for child sleep (CBTcs) to improve sleep in an important high-risk population, overweight/obese (OV/OB) youth with behavioral sleep disorders. OV/OB youth with behavioral sleep disorders and their parent(s) will be randomly assigned to 8 sessions of either CBTcs or an Educational Control (EC). CBTcs will address behavioral sleep issues in children; EC will address sleep and dietary education and general coping strategies. Child sleep (total wake time, total sleep time, bed/wake times), height, weight, physical activity, dietary intake, quality of life (QOL), fatigue, and daytime sleepiness will be assessed at baseline, post-treatment, and 3-month follow-up. It is hypothesized the children in the CBTcs will experience greater improvement in sleep than children in the EC.

DETAILED DESCRIPTION:
Assessment Procedures: Subjects will participate in 8 treatment sessions and 3 full assessment meetings over the course of 7 months. All meetings will be held at the Magnolia Park Sleep Disorders Center. The following procedures will be performed:

Stage 1 - Phone Screening, Stage 2 - Screening and Baseline Measures, Stage 3 - Overnight Sleep Monitoring, Stage 4 - Two weeks Wrist Actigraphy, Sleep Diaries, Dietary Recalls Stage 5 - Intervention, Stage 6 - Post-Treatment Measures, Stage 7 - 3-Month Follow-Up

ELIGIBILITY:
Inclusion Criteria:

* 6-12 years of age
* Prepubescent
* Have a body mass index ≥85th percentile for age and gender norms as published by the CDC, and
* Accompanied by a parent or legal guardian that lives in the same home as the child. The parent must be able to read and understand English at the 5th grade level.

Exclusion Criteria:

* Sleep Apnea: previous diagnosis or an apnea/hypopnea index (AHI) >10 according to PSG.
* Periodic Limb Movement Disorder (PLMD): previous diagnosis or myoclonus arousals per hour >5 according to PSG.
* Circadian Rhythm Sleep Disorder, Delayed Sleep Phase Type
* Medication exclusions: Prescribed or OTC sleep medication within the last 1 month (unless stabilized on medication for 6+ months); Currently taking psychostimulants; antipsychotic agents; monoamine oxidase inhibitors; systemic corticosteroids; antibiotics for HIV or TB; chemotherapeutic drugs; or use of prescription weight-loss drugs within six months.
* Conditions or behaviors likely to affect trial conduct: unwilling to accept random assignment; participation in another randomized research project; parent unable to read and understand English at the 5th grade level; presence of bipolar or seizure disorder (potential sleep restriction); restless leg syndrome, major psychiatric disorder other than anxiety or depression; child with major cognitive or developmental delay; unable to complete forms, implement treatment procedures, etc. due to cognitive impairment; psychotropic or other medications (beta-blockers) known to alter sleep; participation in other CBT treatment or nonpharmacological sleep treatment; or any other condition/situation which would adversely affect trial participation.

Ages: 6 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 54 (Actual)
Dates: Start 2014-09 (Actual); Primary Completion 2017-08-30 (Actual); Study Completion 2017-09-30 (Actual)

PRIMARY OUTCOMES:
Total Sleep Time | change from baseline to 2 months

SECONDARY OUTCOMES:
time spent in physical activity | change from baseline to 2 months
caloric intake | change from baseline to 2 months

CONTACTS AND LOCATIONS:
Overall Officials: David M Janicke, PhD, Principal Investigator — University of Florida; Christina McCrae, PhD, Principal Investigator — University of Florida
Locations (1):
- UF Health Shands, Gainesville, Florida, United States